CLINICAL TRIAL: NCT03524365
Title: A Randomized Controlled Study on the Effects of Roux-en-Y Gastric Bypass Versus Sleeve Gastrectomy or Intensive Lifestyle Modifications on Non Alcoholic Steato-Hepatitis
Brief Title: Bariatric Surgery Versus Non-alcoholic Steato-hepatitis
Acronym: BRAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Associate Professor of Internal Medicine, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20182004
Record Dates: First submitted 2018-04-21; First posted 2018-05-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RYGB plus LM counselling (Active Comparator): 96 subjects with NASH
  Interventions: Procedure: RYGB
- SG plus LM counselling (Active Comparator): 96 subjects with NASH
  Interventions: Procedure: SG
- ILM (Sham Comparator): 96 subjects with NASH
  Interventions: Other: Intensive Lifestyle Modification

INTERVENTIONS:
Procedure: RYGB — Roux-&-Y Gastric Bypass (RYGB) involves the use of a surgical stapler to create a small and vertically oriented gastric pouch with a volume of 30 ml. The upper pouch is completely divided by the gastric remnant and is anastomosed to the jejunum, 75 cm distally to the Treitz's ligament , through a narrow gastrojejunal anastomosis in a Roux-en-Y fashion. Bowel continuity is restored by an entero-entero anastomosis, between the excluded biliary limb and the alimentary limb, performed at 100 cm from the gastrojejunostomy. Lifestyle modification counselling is provided to each patient.
  Arms: RYGB plus LM counselling
Procedure: SG — The SG is created using a linear stapler with two sequential 4.8/60-mm green load firings for the antrum, followed by two or three sequential 3.5/60-mm blue loads for the remaining gastric corpus and fundus. The stapler is applied alongside a 48-Fr calibrating bougie. The resection line is performed avoiding the ''critical area'' by resecting the fundus 1.5 cm from the angle of His. Staple lines are buttressed with bovine pericardial strips. The resected stomach is grasped at the antral tip by a laparoscopic grasper and retrieved through one of the trocar sites. A methylene blue dye test by a nasogastric tube is routinely performed at the end of the procedure. The residual gastric remnant capacity is 60-80 ml. Drains are not routinely placed, and the nasogastric tube is removed at the end of the procedure. Upper gastrointestinal contrast (Gastrografin) study is performed on the first postoperative day. Lifestyle modification counselling is provided to each patient.
  Arms: SG plus LM counselling
Other: Intensive Lifestyle Modification — Resting calorie requirements will be calculated via the Harris Benedict equation (24) and an activity factor, and subjects will be instructed not to change their activity level other than that suggested by physicians during the study. The diet will contain 1/3 kcal less than the calculated energy expenditure and 30% fat of which 10% saturated, 55% lower glycemic index carbohydrates and 15% proteins.
  The participants will be encouraged to gradually increase their walking to achieve 10,000 steps per day. A moderate intensity physical activity program of 1 hour of aerobic exercise 2-3 hours per week will be recommended to all subjects. Their physical activity will be assessed by IPAQ-SF.
  Arms: ILM

SUMMARY:
Bariatric-metabolic surgery is effective in treating the cluster of conditions forming the metabolic syndrome, strictly associated with NAFLD and NASH. Recently, we and other authors have shown also in the long term (up 5 years) with randomized-controlled trials (RCTs) that bariatric-metabolic surgery allows remission of type 2 diabetes and obesity reduction, which are the two major pathogenetic factors of NASH development, with maintenance of weight loss.

Few small and mainly retrospective studies have shown that bariatric surgery is effective in improving NASH histologic picture in obese subjects.

The aim of our proposal is to conduct a 3 arm single centre, superiority, RCT comparing Roux-en-Y Gastric Bypass (RYGB) with Sleeve Gastrectomy (SG) and with Intensive Lifestyle Modifications (ILM) for the treatment of Non-Alcoholic Steato-Hepatitis.

DETAILED DESCRIPTION:
This is a Randomized Controlled multicentre Trial involving the Catholic University (Professor Geltrude Mingrone as PI and Professor Marco Raffaelli as co-PI)

The research question in PICOT format (P) - Population: Adults 25 to 70 years of age and BMI ≥ 30 and ≤55 kg/m2 with histological diagnosis of NASH.

(I) - Intervention: Roux-en-Y Gastric Bypass or Sleeve Gastrectomy, both plus lifestyle counseling.

(C) - Comparison: Intensive Lifestyle Modifications. (O) - Outcome: the histological resolution of NASH without worsening of fibrosis at 1 year after the interventions.

(T) - Time: One year after the intervention started.

1.3.3.2 Research Goals

* The primary aim of our study is to assess the effects of bariatric-metabolic surgery or ILM on NASH at 1 year after the interventions.
* Secondary aims are to assess the safety of bariatric surgery and the improvement of at least 1 stage of liver fibrosis without worsening of NASH, insulin sensitivity , T2DM, and lipoprotein profile changes.

The liver biopsy will be performed at baseline and at 1 year follow-up. Another liver biopsy will be performed at 3 and 5 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with NASH documented by liver biopsy and no evidence of another form of liver disease with a BMI ≥ 30 and ≤55 kg/m2.

Subjects with normal liver who underwent laparoscopic elective cholecystectomy, but otherwise in healthy conditions, will be used as controls for the discovery of non-invasive biomarkers.

Exclusion Criteria:

* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous 6 months; Liver cirrhosis; End stage renal failure; Participation in any other concurrent therapeutic clinical trial; Any other life-threatening, non-cardiac disease; Pregnancy; Inability to give informed consent; Substantial alcohol consumption (>20 g/day for women or >30 g/day for men); Wilson's disease;hepatitis B virus, hepatitis C virus (negative Hepatitis C RNA since more than 3 years will be considered eligible), autoimmune hepatitis, primary biliary cholangitis, haemochromatosis and α-1-antitrypsin deficiency; Lipodystrophy; Parenteral nutrition; Abetalipoproteinemia; Interfering medications (e.g., amiodarone, methotrexate, tamoxifen, corticosteroids).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
histological resolution of NASH without worsening of fibrosis at 1 year after the interventions | 1 year
  Histological diagnosis of NASH is established according to widely accepted criteria, using the NAFLD activity score (NAS) algorithm proposed by the NASH Clinical Research Network (CRN). These criteria include presence of steatosis in >5% of hepatocytes, hepatocellular ballooning and lobular inflammatory infiltrates. The presence and stages of fibrosis will be also assessed using the NASH-CRN system: stage 0 =no fibrosis; stage 1 =centrilobular pericellular fibrosis; stage 2 =centrilobular and periportal fibrosis; stage 3 =bridging fibrosis; and stage 4 =cirrhosis.

SECONDARY OUTCOMES:
Adverse health events including the need for re-operation | 1 year
  adverse events include early operation complications
Improvement of at least 1 point of histological liver fibrosis without worsening of NASH | 1 year
  liver fibrosis will be examined in liver biopsies
Changes in glycemic control (only in diabetic patients) | 1 year
  diabetes remission or improvement of glycemic control (glycated hemoglobin HbA1c)
Changes in insulin sensitivity | 1 year
  HOMA IR or oral glucose minimal model
Changes in food intake | 1 year
  food intake diary
Changes in physical activity | 1 year
  Physical activity questionnaire
Changes in body composition: Fat-Free Mass (FFM), Fat Mass (FM). | 1 year
  FFM and FM will be assessed by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD PhD, Principal Investigator — Catholic University
Locations (3):
- Italy (3):
  - San Camillo, Roma
  - University of Rome Sapienza, Roma
  - Catholic University School of Medicine, Rome

REFERENCES:
- [Derived] Angelini G, Panunzi S, Pompili M, Riccardi L, Garcovich M, Verrastro O, Russo S, Mare T, Luxton J, le Roux CW, Raffaelli M, Mingrone G, Vincent RP. Performance of Noninvasive Tests for Metabolic Dysfunction-Associated Steatohepatitis and Liver Fibrosis Resolution after Bariatric Surgery. Clin Chem. 2025 Mar 3;71(3):406-417. doi: 10.1093/clinchem/hvae208. PMID 39786442
- [Derived] Verrastro O, Panunzi S, Castagneto-Gissey L, De Gaetano A, Lembo E, Capristo E, Guidone C, Angelini G, Pennestri F, Sessa L, Vecchio FM, Riccardi L, Zocco MA, Boskoski I, Casella-Mariolo JR, Marini P, Pompili M, Casella G, Fiori E, Rubino F, Bornstein SR, Raffaelli M, Mingrone G. Bariatric-metabolic surgery versus lifestyle intervention plus best medical care in non-alcoholic steatohepatitis (BRAVES): a multicentre, open-label, randomised trial. Lancet. 2023 May 27;401(10390):1786-1797. doi: 10.1016/S0140-6736(23)00634-7. Epub 2023 Apr 21. PMID 37088093
- [Derived] Angelini G, Panunzi S, Castagneto-Gissey L, Pellicano F, De Gaetano A, Pompili M, Riccardi L, Garcovich M, Raffaelli M, Ciccoritti L, Verrastro O, Russo MF, Vecchio FM, Casella G, Casella-Mariolo J, Papa L, Marini PL, Rubino F, le Roux CW, Bornstein S, Mingrone G. Accurate liquid biopsy for the diagnosis of non-alcoholic steatohepatitis and liver fibrosis. Gut. 2023 Feb;72(2):392-403. doi: 10.1136/gutjnl-2022-327498. Epub 2022 Jul 12. PMID 35820779